CLINICAL TRIAL: NCT01719328
Title: The Effects of Vinayasa Yoga on Mood and Stress
Brief Title: Vinayasa Yoga and Mood
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Responsible Party: Principal Investigator, Beth Bock, Ph.D., Professor of Psychiatry and Human Behavior, The Miriam Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R21AT003669-01S1 (NIH)
Record Dates: First submitted 2012-10-30; First posted 2012-11-01 (Estimated); Last update posted 2013-10-24 (Estimated); Status verified 2013-10

CONDITIONS: Affect; Stress, Psychological
Keywords: yoga,; exercise; affect; mind/body therapies; stress, psychological
MeSH Terms: conditions — Stress, Psychological; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vinyasa yoga (Experimental): Group administered 60 minute vinyasa yoga classes delivered twice weekly for 8 weeks
  Interventions: Behavioral: Vinyasa yoga

INTERVENTIONS:
Behavioral: Vinyasa yoga

SUMMARY:
The purpose of this study is to examine the immediate and cumulative effects of yoga on stress and mood among young adult college students attending an 8-week program in Vinyasa yoga.

DETAILED DESCRIPTION:
Traditional vigorous aerobic exercises (TAE), such as running and bicycling have been shown to improve mood and relieve stress. Yoga is an ancient physical and mental practice that as a form of exercise may share properties of TAE and in turn offer similar mood and stress effects. However, scientifically rigorous studies examining the psychological effects of yoga and published in peer-reviewed Western journals are rare. The aim of this research was to establish preliminary evidence for the acute effects of vinyasa yoga on mood and stress among young adults.

ELIGIBILITY:
Inclusion Criteria:

* Adult ages 18 or older
* English-speaking

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2007-02; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beth C Bock, PhD, Principal Investigator — Brown Alpert Medical School, The Miriam Hospital
Locations (1):
- The Miriam Hospital- CORO building, Providence, Rhode Island, United States